CLINICAL TRIAL: NCT01274403
Title: A Randomized Study With Oral Melphalan + Prednisone (MP) Versus Melphalan, + Prednisone + Thalidomide (MPT) for Newly Diagnosesd Elderly Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Studio Linfomi (Other)
Responsible Party: Gruppo Italiano Studio Linfoma, GISL
Allocation: Randomized | Masking: None
Other Study IDs: MM03
Record Dates: First submitted 2010-12-28; First posted 2011-01-11 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2010-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Elderly patients
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Prednisone; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melphalan, prednisone plus Thalidomide (Experimental)
  Interventions: Drug: Melphalan, Prednisone and Thalidomide
- Melphalan and Prednisone (Active Comparator)
  Interventions: Drug: Melphalan, Prednisone and Thalidomide

INTERVENTIONS:
Drug: Melphalan, Prednisone and Thalidomide

SUMMARY:
The aim of the study is to compare efficacy and toxicity of melphalan and prednisone versus meplhalan, prednisone and Thalidomide in elderly patients with multiple myeloma or patients with multiple myeloma but not eligible for high dose treatment with stem cells support.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed of multiple myeloma.
* Age > 65 years
* ECOG <= 3
* Written informed consent given at the time of randomization
* Patients with age <= 65 but not eligible for high dose treatment with stem cells support

Exclusion Criteria:

* ECOG > 3
* current neoplasm..
* contraindications to use thalidomide
* peripheral neurophaty

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 130 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy | from 8 to 12 months
  To compare the percentage of response in term of complete response, partial response, minimal and stable disease in the 2 arms o treatment
To assess the toxicity | From 1 to 12 months
  To evaluate the toxicity in the 2 arms of treatment utilized the common terminology criteria for adverse events (CTCAE) version 3.0

SECONDARY OUTCOMES:
To evaluate the Overall Survival (OS) in the 2 arms of treatment | From 1 to 60 months
  OS was defined as the time from the date of first treatment after diagnosis of multiple myeloma to the date of last follow up examination or the date of death from any cause
To evaluate the Duration of Remission (DR) in the 2 arms of treatment | From 8 to 60 months
  DR was defined from the date of Complete Remission, Partial Remission, Minimal response after the completion of MPT or MP cycles to the date of disease progression or the date of last follow up examination

CONTACTS AND LOCATIONS:
Locations (1):
- Gruppo Italiano Studio Linfoma, Modena, Modena, Italy